CLINICAL TRIAL: NCT06245122
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of CS23546 in Subjects With Advanced Tumors
Brief Title: A Study of CS23546 in Subjects With Advanced Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CS23546-101
Record Dates: First submitted 2023-12-26; First posted 2024-02-07 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Advanced Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose escalation (Experimental): Single ascending dose (SAD): Participants will receive CS23546 once on the first day (D1).
  Multiple ascending dose (MAD): Participants will receive CS23546 once daily from the 7th day (C1D1).
  Interventions: Drug: CS23546
- Dose expansion (Experimental): Dose expansion is planned to begin when the recommended Phase 2 dose (RP2D) will be determined.
  Interventions: Drug: CS23546

INTERVENTIONS:
Drug: CS23546 — Tablets administered orally.

SUMMARY:
The primary objectives of this study are to characterize the safety and tolerability of CS23546 and to evaluate the pharmacokinetic (PK) characteristics and recommended phase 2 dose (RP2D) of CS23546 in subjects with advanced tumors.

DETAILED DESCRIPTION:
This study is a single arm, open phase I trial, consisting of a dose escalation phase (single dose+multiple doses) and a dose expansion phase, accompanied by pharmacokinetic and pharmacokinetic studies. The first visit period (21 days) of single dose and multiple doses during the dose-increasing phase is the DLT observation period.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female and ≥18 years of age on day of signing informed consent.
2. Histologically or cytologically confirmed unresectable advanced recurrent/refractory solid tumor or lymphoma that is failure or or intolerant of all standard therapy or for which no standard therapy is available.
3. Individuals are required to provide tumor tissue samples for prospective detection of Programmed cell death 1 ligand 1 (PD-L1) expression and/or Microsatellite instability (MSI) / the DNA mismatch repair (MMR) status. Subjects who cannot be provided during the dose escalation phase will be evaluated by the researchers and sponsors before deciding whether to enroll.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
5. Adequate organ function.
6. Life expectancy ≥12 weeks.
7. Dose expansion phase: Cohort 1, Subjects with urothelial carcinoma. Cohort 2, Subjects with Extranodal NK/T-cell lymphoma (NKTCL). Cohort 3, Subjects with soft tissue sarcoma. Cohort 4, Subjects with PD-L1 expression positive and/or microsatellite-instability-high (MSI-H) / mismatch-repair-deficient (dMMR) advanced solid tumors or lymphoma

Key Exclusion Criteria:

1. Received anti-tumor therapy (including but not limited to chemotherapy, targeted therapy, anti angiogenic therapy, immunotherapy, cell therapy, radiotherapy, tumor embolization, etc.) or experimental drugs/devices that have not been approved for marketing within 28 days before the first medication.
2. History of ≥ Grade 3 immune related Adverse Events (irAEs) or termination of treatment due to irAEs during prior treatment with Programmed death 1 (PD-1) /PD-L1 antibody.
3. Active autoimmune diseases present during the screening period and systemic treatment was received within 2 years before the first medication. Individuals who only require hormone replacement therapy (such as thyroxine, insulin, or physiological corticosteroids used for adrenal or pituitary insufficiency) can be enrolled.
4. Presence of central nervous system metastasis and/or meningeal metastasis.
5. Dose expansion phase: Subjects with solid tumors or lymphoma who have previously received PD-L1 inhibitors and belong to primary resistance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLTs) | Day 1 through Day 27
  DLT: Number of patients experienced any dose limited toxicity. MTD: One level lower than the dose level at which dose escalation was terminated due to DLT reasons.
Maximum Tolerated Dose (MTD) | Day 1 through Day 27
  MTD: One level lower than the dose level at which dose escalation was terminated due to DLT reasons.
Time to Cmax (Tmax) | up to Day 1 of cycle 5 (each cycle is 21 days)
  Time to reach the Cmax for CS23546.
Maximum plasma concentration (Cmax) | up to Day 1 of cycle 5 (each cycle is 21 days)
  Maximum observed plasma concentration for CS23546.
Area Under the Curve (AUC) | up to Day 1 of cycle 5 (each cycle is 21 days)
  Area Under the Plasma Concentration-time Curve From Zero Time to the Last Measurable Point for CS23546.

SECONDARY OUTCOMES:
The inhibitory activity of Programmed cell death 1 ligand 1 (PD-L1) | up to Day 1 of cycle 5 (each cycle is 21 days)
Interferon gamma (IFN-γ) | up to Day 1 of cycle 5 (each cycle is 21 days)
  Plasma concentration for IFN-γ.
Free PD-L1 | up to Day 1 of cycle 5 (each cycle is 21 days)
  Plasma concentration for free PD-L1.
C-X-C motif chemokine 9 (CXCL9) | up to Day 1 of cycle 5 (each cycle is 21 days)
  Plasma concentration for CXCL9.
C-X-C motif chemokine 10 (CXCL10) | up to Day 1 of cycle 5 (each cycle is 21 days)
  Plasma concentration for CXCL10.
Objective response rate (ORR) | Until 28 days after the last dose of the study drug
  Efficacy evaluation indicators for research.
Disease control rate (DCR) | Until 28 days after the last dose of the study drug
  Efficacy evaluation indicators for research.
Duration of response (DOR) | Until 28 days after the last dose of the study drug
  Efficacy evaluation indicators for research.
Time to progression (TTP) | Until 28 days after the last dose of the study drug
  Efficacy evaluation indicators for research.
time to progressive disease (TTR) | Until 28 days after the last dose of the study drug
  Efficacy evaluation indicators for research.
Progression free survival (PFS) | Until 28 days after the last dose of the study drug
  Efficacy evaluation indicators for research.
Overall survival (OS) | Until 28 days after the last dose of the study drug
  Efficacy evaluation indicators for research.
Safety indicators: adverse events (AE) | Until 28 days after the last dose of the study drug
  The incidence and severity of adverse events (AE) (according to CTCAE v5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Huiqiang Huang, Ph.D., Principal Investigator — Sun Yat-sen University Cancer Cancer
Locations (1):
- Sun Yat-sen University Cancer Cancer, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No